CLINICAL TRIAL: NCT04068675
Title: Effects of Centering Pre-operative Counseling on Patient Reported Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Emma Barber, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00209941
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Gynecologic Cancer; Ovarian Cancer; Endometrial Cancer; Uterine Cancer; Cervical Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group counseling arm (Experimental): There is only one(1) arm in this study. All patients that enroll in the study will receive the group counseling intervention and be compared to historical controls.
  Interventions: Behavioral: Group pre-operative counseling

INTERVENTIONS:
Behavioral: Group pre-operative counseling — Enrolled patients will participate in a group pre-operative counseling session on the online conferencing platform BlueJeans® prior to their surgery. The sessions will not replace any portion of the pre-operative standard counseling and is designed to review and re-enforce the counseling already provided. The sessions will not review or discuss the specifics of any one individual's cancer or surgery. Rather the counseling session will focus on the universal instructions provided to all patients undergoing major surgery for a known or suspected gynecologic malignancy. The sessions will be led by a physician on a weekly basis with a minimal of three (3) enrolled patients per session and last approximately one (1) hour.

SUMMARY:
The primary objective of the study is to evaluate the effect of pre-operative counseling in a group setting on patient reported anxiety for patients scheduled to undergo surgery for a known or suspected gynecologic malignancy. Patient reported anxiety will be evaluated using a validated Patient-Reported Outcomes Measurement Information System (PROMIS) survey. We hypothesize that the group counseling session will reduce patient reported anxiety by a clinical meaningful level. Secondary objectives will evaluate the effect of the intervention on patient reported depression levels and compare adherence to Enhanced Recovery After Surgery (ERAS) instructions, utilization of unscheduled health care resources, and anxiety/depression levels to historical controls.

DETAILED DESCRIPTION:
Comprehensive pre-operative counseling and education has been shown to play an important role in quality of life, anxiety and depression among cancer patients. Traditionally, patients are counseled in the office at the time of informed surgical consent. However there are several problems to this model including patient anxiety, confusion, information overload, and time constraints that may lead to sub-optimal counseling. Additionally, multiple studies have reported that patients forget half of what they have been told within 5 minutes of a health consultation and remember only 20% of the information passed on to them. Centering patient counseling has been used in other fields of medicine and has been shown to improve outcome in Obstetrics, Psychiatry, Gastroenterology, and Medical Oncology. In Obstetrics, centering pre-natal care with group counseling sessions has shown to be an effective model for improving perinatal outcomes and patient satisfaction. Pregnancy, not unlike cancer, is a medical condition that rapidly change's one life, is marred by anxiety, nervousness and innumerable potential symptoms. The rationale behind centering care is that providers can spend more time counseling and educating a larger audience at once, and it allows the whole group to benefit from individual questions, concerns, and complaints. Additionally, it establishes a network for patients to connect with other women going through similar stressors.

Prior to initiating this study, we conducted an Institutional Review Board exempt survey (STU00209351) of patients scheduled to undergo surgery with one of our Gynecologic Oncologists. Over 68% of patients expressed an interest in participating in a study to receive additional counseling. However, re-occurring themes that were mentioned were the time constraints and commuting issues in which patients experience in coming to our clinic in downtown Chicago. Given this feedback and the strong interest that our patient population has for this type of intervention, we have modified the traditional in-person centering model to an internet base, video conference group counseling session.

ELIGIBILITY:
Inclusion Criteria:

* Women equal to or greater than 18 years old
* Fluent in English
* Known or suspected diagnosis of a gynecologic malignancy (ovarian, endometrial, uterine, and cervical cancers)
* Scheduled for major surgery at Northwestern Memorial Hospital/Prentice Women's Hospital (any laparotomy or laparoscopic or robotic assisted hysterectomy) within 4 weeks of study enrollment
* Internet access and ability to complete online survey and online counseling session

Exclusion Criteria:

* Under 18 years of age
* Adults unable to consent (cognitive impairment)
* Pregnant women
* Prisoners
* Urgent/Emergent surgery (surgery in less than 72 hours of consultation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have a known or suspected gynecologic malignancy to be eligible for this study
Enrollment: 75 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety survey scores | It will take no more than 8 weeks to complete all survey related activities.
  The PROMIS Anxiety survey is a validated survey tool used to measure the severity of patient reported anxiety. Responses from the survey are converted to a T-score (scale: minimum score = 37.1, maximum score = 83.1) which have been standardized to the US general population with a mean 50 and standard deviation of 10. A score of less than 50 correlates to "normal" levels of anxiety, where as a score of 50-60 represents mild anxiety, 60-70 represents moderate anxiety, and >70 represents severe anxiety. PROMIS Anxiety scores will be evaluated at time of enrollment, after receiving the intervention, and four (4) weeks after surgery to evaluate for changes in anxiety scores.

SECONDARY OUTCOMES:
Changes in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression survey scores | It will take no more than 8 weeks to complete all survey related activities.
  The PROMIS Depression survey is a validated survey tool used to measure the severity of patient reported depression. Responses from the survey are converted to a T-score (scale: minimum score = 37.1, maximum score = 83.1) which have been standardized to the US general population with a mean 50 and standard deviation of 10. A score of less than 50 correlates to "normal" levels of depression, where as a score of 50-60 represents mild depression, 60-70 represents moderate depression, and >70 represents severe depression. PROMIS Depression scores will be evaluated at time of enrollment, after receiving the intervention, and four (4) weeks after surgery to evaluate for changes in depression scores.
Hospital length of stay | From surgery through study completion, an average of 4 weeks.
  The number of total days spent in the hospital after surgery until discharge
Enhanced Recovery After Surgery (ERAS) compliance | From surgery through study completion, an average of 4 weeks.
  Compliance with ERAS instructions
Unscheduled health care resource use in the post-operative period | From surgery through study completion, an average of 4 weeks.
  Use of unscheduled health care resources such as hospital re-admissions, ER visits, unscheduled clinic visits, problem-related phone calls and emails after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barber, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No